CLINICAL TRIAL: NCT04412954
Title: Improving Cardiovascular Risk Factors in Black Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Janna Stephens, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2019B0560
Record Dates: First submitted 2020-05-18; First posted 2020-06-02 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Obesity
Keywords: minority; College Student; Nutrition; Physical Activity; Health Coach
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Health coach with Smartphone application for diet and physical activity
  Interventions: Behavioral: Smartphone + Text Messaging with Health Coach
- Control (No Intervention): No intervention, using a Smartphone application for sleep monitoring

INTERVENTIONS:
Behavioral: Smartphone + Text Messaging with Health Coach — The program includes (1) use of a free commercially available smartphone application program for 12 months, (2) a wearable Fitbit Charge device that will be provided by the study to monitor active minutes, and (3) one 45-minute behavioral counseling session focused on healthy eating and exercise and (4) personalized text messaging for 6 months by a health coach. The health coach will not send feedback during months 6-12. The intervention will be fully self-directed in these months, as there will be no contact between the 6 months visit and 12-month visit.
  Arms: Intervention

SUMMARY:
The objectives of the study are to conduct a randomized controlled trial to test the efficacy of the Smartphone intervention on % weight loss and maintaining % weight loss at 6 and 12 months in a sample (N=256) of Black community college students who are overweight or obese, ages 18-25 years. Investigators will also examine mediating variables of the intervention on weight at 6 and 12 months, including adherence to self-monitoring, discrimination, and dietary and physical activity self-efficacy. In addition, investigators will explore potential moderators of weight loss at 6 months and 12 months, including depressive symptoms, ideal body image, and motivation.

DETAILED DESCRIPTION:
A total of 256 students, ages 18-25, who meet the inclusion and exclusion criteria will be recruited from Columbus State Community College (CSCC). A sample size of 256 subjects (n=128 per each trial arm) will have sufficient power (>80%) to detect an average between-group difference with a moderate effect size of 0.4. The mixed effect modeling for repeated outcome measures at 6 and 12 months was used for the power calculation using two-sided significance level of 0.05 assuming 1) first-order autoregressive covariance structure, 2) the within-structure correlation of 0.8, and 3) 20% attrition rate at 12-month follow-up. The effect size of 0.4 was reasonably assumed based on data from published trials on weight-loss interventions (an effect size of 0.8 using 8-week social media, 0.3 using 12-week Smartphone intervention, and 0.6 using 4-month text messaging). Investigators will conduct stratified recruitment by gender (female vs. male) and ethnicity (Non-Hispanic Black vs. Hispanic Black) to achieve a study sample with 80% Non-Hispanic Black and 20% Hispanic and 50% male in each ethnic group. The recruitment and randomization will be equally distributed with approximately 10 subjects per month, which is a feasible enrollment target considering the pool of eligible participants and our previous recruitment success.

Prospective participants who contact through telephone or email will undergo a preliminary screening via telephone and receive an explanation of the study. Included in this screening are four questions from the Eating Attitude Test-26 (EAT-26), which will be asked to determine symptoms of disordered eating in the past 6 months. Those who seem to meet eligibility criteria and are interested in participating will be scheduled for an in person visit for the informed consent and screening process.

Following the informed consent process and baseline visit questionnaires, participants will be randomly assigned to intervention or the attention-control group. Investigators will use stratified randomization by sex (female vs. male) and ethnicity (Non-Hispanic Black vs. Hispanic Black). For each gender strata, randomization will occur in permuted blocks of varying block sizes. Subjects in each block will be randomly assigned to intervention arm or attention-control arm with an allocation ratio of 1:1. The advantage of permuted block randomization is that it will ensure balance in the number of subjects in the two trial arms during the entire study period.

ELIGIBILITY:
Inclusion

* age 17-25 years
* Current CSCC student
* Identify as Black
* BMI ≥ 25
* Speaks and reads English
* Interested in losing weight through diet and physical activity changes
* Owns a smartphone or iPhone Operating System (iOS) or Android compatible device
* Ability to return for 12-month visit

Exclusion

* currently pregnant or planning to become pregnant in next 12 months
* Currently participating in another structured weight loss program or taking weight loss medications or medication known to increase weight
* Lost 10% or more of body weight in past 6 months
* Screens positive for disordered eating symptoms
* diagnosed with type I diabetes

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 256 (Actual)
Dates: Start 2020-12-05 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stephens J, Randolph J, Burke L, Miller C, Tan A, Buffington B, Melnyk B, Perkins A. A randomized controlled trial for reduction of risk factors for cardiovascular disease in young adults: Methods of the Aspire study. Contemp Clin Trials. 2022 Oct;121:106873. doi: 10.1016/j.cct.2022.106873. Epub 2022 Sep 5. PMID 36070664
- [Derived] Leissa SM, Randolph JC, Stephens JD. Recruitment of Black Identifying Young Adults into Clinical Trials: a Report from the Field. J Urban Health. 2021 Oct;98(Suppl 2):155-159. doi: 10.1007/s11524-021-00569-4. Epub 2021 Aug 13. No abstract available. PMID 34389927

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 128 | 128
Completed | 98 | 108
Not Completed | 30 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 128 | 128 | 256
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 126 | 126 | 252
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 64 | 128
  Male | 64 | 64 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 23 | 45
  Not Hispanic or Latino | 106 | 105 | 211
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 90 | 92 | 182
  White | 0 | 0 | 0
  More than one race | 38 | 36 | 74
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 128 | 128 | 256
Weight [Mean (Standard Deviation); unit: Pounds] | 208.9 (49.2) | 210.6 (43.9) | 209.4 (45.6)
Body Mass Index [Mean (Standard Deviation); unit: weight (lb) ÷ height2 (inches) * 703] | 32.8 (7.1) | 33.3 (6.0) | 33.2 (6.4)
Active Minutes Exercise [Mean (Standard Deviation); unit: Minutes] | 30.5 (40.4) | 27.2 (37.8) | 28.9 (39.1)
Steps Exercise [Mean (Standard Deviation); unit: Steps per day] | 5553 (4274) | 5452 (4289) | 5503 (4281)
Patient Health Questionnaire 9 [Mean (Standard Deviation); unit: Score on a scale] — This is the patient health questionnaire 9 survey. Total score is reported. Scale ranges from 0-27. Higher values represents more depressive symptoms, thus we want to see lower scores.
  Score on a scale | 6.5 (4.8) | 6.6 (4.8) | 6.6 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: Body weight will be measured in light clothing without shoes using the Tanita Body Scale (BS)
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: Pounds
Groups:
- Control: Control condition received an application for sleep
- Intervention: Intervention group received health coaching and a smartphone application for weight loss.
Arm/Group | Control | Intervention
Number analyzed (Participants) | 108 | 108
Pounds | -2.5 (15.3) | -0.8 (17.2)

2. Primary Outcome: Physical Activity-Active Minutes/Day
Description: Will be measured objectively using the FitBit Charge for 7 days at each time period of data collection. Average active minutes per day will be used as measurement. This data represents active minutes per day at 12 months
Time Frame: 12 months
Population: minutes/day
Measure: Mean (Standard Deviation); unit: Minutes/day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 98 | 103
Minutes/day | 9.7 (21) | 12.9 (24.2)

3. Primary Outcome: Physical Activity-Steps/Day
Description: Will be measured objectively using the FitBit Charge for 7 days at each time period of data collection. Average steps taken per day will be used as measurement.
Time Frame: 12 months
Population: steps/day
Measure: Mean (Standard Deviation); unit: Steps/day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 95 | 99
Steps/day | 2537 (4333) | 2659 (3853)

4. Primary Outcome: Food Frequency Questionnaire (FFQ)
Description: The full-length block FFQ will be used to assess diet for 7 days at each period of data collection. This is not a scale, this is a measure of foods consumed over a period of 7 days. We measured and target sodium as the nutrient of choice to analyze
Time Frame: 12 months
Population: mg of sodium/day
Measure: Mean (Standard Deviation); unit: Mg of sodium per day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 110 | 105
Mg of sodium per day | 3503 (1205) | 4105 (1100)

5. Primary Outcome: Healthy Eating Index (HEI)
Description: A healthy eating index score will be calculated at each time period from the FFQ. The scale ranges from 0-100 with 100 being the best possible score indicating healthy diet aligning with key dietary recommendations.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 110 | 105
Score on a scale | 47 (6.8) | 48 (7.1)

6. Secondary Outcome: Rate of Participants Who Are Adherent to Self-Monitoring
Description: Intervention condition only. Adherence will be defined as those participants who enter at least 50% of their caloric goal on at least 80% of days (or 24 days per months).
Time Frame: Baseline to 12 months
Population: Intervention group who used app on or more than 80% of days to enter food
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 124
Participants | 40

7. Secondary Outcome: Dietary Self-Efficacy Scale (Diet-SE)
Description: 14 questions that examine the participant's belief in their ability to cut down on high caloric foods. Scale ranges from 0-4 with 0 being "not at all confident" and 4 being "very confident" Higher overall score indicates higher levels of self confidence. Total score ranges from 0-56. Total score is reported.
Time Frame: 12 months
Population: 12 month total score
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 97 | 98
score on a scale | 27.8 (9.7) | 25.4 (10.1)

8. Secondary Outcome: Self-Efficacy for Exercise Scale
Description: 9 questions that examine the participant's belief in their ability to complete physical activity in given circumstances. Scale ranges from 0-10 with 0 being not at all confident and 10 being the most confident. Overall scores range from 0-90 with 90 indicating high confidence levels for exercise.
Time Frame: 12 months
Population: Total score at 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 97 | 98
score on a scale | 48.9 (22.2) | 50.1 (23.2)

9. Secondary Outcome: Experiences of Discrimination Scale (EoD)
Description: Examines perceived experiences of discrimination in given circumstances, such as work, public settings, banks, schools, medical care. 17 questions total. Scale ranges from never to four or more times. Four or more times being selected indicates higher levels of discrimination experiences. Total score reported. Higher score means higher levels of discrimination. Total score can range from 0 - 68
Time Frame: 12 months
Population: Total score at 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 107 | 113
score on a scale | 8.8 (9.5) | 9.3 (9.5)

10. Secondary Outcome: Patient Health Questionnaire (PHQ) for Adults, PHQ-9
Description: Measures depressive symptoms using the patient health questionnaire for adults. Questions are scored from 0-3, with lower scores indicating no/lower depressive symptoms. Total score can range from 0-27
Time Frame: 12 months
Population: Total score at 12 months
Measure: Mean (Standard Deviation); unit: Total score on scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 97 | 98
Total score on scale | 5.8 (4.9) | 5.5 (4.2)

11. Secondary Outcome: Ideal Body Image
Description: Measures patient perception of their current body image and their ideal body. image using a graphic scale ranging from 0-9, with 9 indicating higher levels of overweight/obesity.
Time Frame: 12 months
Population: Ideal body image at 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention Female; Intervention Male: Health coach with Smartphone application for diet and physical activity
  Smartphone + Text Messaging with Health Coach: The program includes (1) use of a free commercially available smartphone application program for 12 months, (2) a wearable Fitbit Charge device that will be provided by the study to monitor active minutes, and (3) one 45-minute behavioral counseling session focused on healthy eating and exercise and (4) personalized text messaging for 6 months by a health coach. The health coach will not send feedback during months 6-12. The intervention will be fully self-directed in these months, as there will be no contact between the 6 months visit and 12-month visit.
- Control Female; Control Male: No intervention, using a Smartphone application for sleep monitoring
Arm/Group | Intervention Female | Control Female | Intervention Male | Control Male
Number analyzed (Participants) | 51 | 50 | 43 | 48
score on a scale | 3.9 (1.1) | 3.5 (0.9) | 4.1 (1.2) | 3.9 (0.9)

12. Secondary Outcome: Treatment Self-Regulation Questionnaire (TSRQ) for Diet and Exercise
Description: 30 questions to measure motivation to lose weight by examining three types of motivation. Scale ranges from 0-7 with 0 being "not at all" and 7 being "very true". A higher score indicates higher levels of motivation for diet and exercise habits. Total score can range from 0 - 210
Time Frame: 12 months
Population: Score at 12 months
Measure: Mean (Standard Deviation); unit: Score on survey
Arm/Group | Intervention | Control
Number analyzed (Participants) | 97 | 98
Score on survey | 59.7 (11.3) | 61.2 (12.7)

13. Secondary Outcome: NIH Patient Reported Outcome Measurement Information System (PROMIS) Measure for Emotional Support
Description: 16 questions to measure perceived levels of emotional support. Scale ranges from 1-5 with 1 being "never" and 5 being "always. A higher level score indicates higher level of emotional support. Total scores can range from 16-80
Time Frame: 12 months
Population: Total Score at 12 months
Measure: Mean (Standard Deviation); unit: Score on survey
Arm/Group | Intervention | Control
Number analyzed (Participants) | 97 | 98
Score on survey | 63 (13.8) | 64.2 (15.0)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of the participant's time in the study, 12 months.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/128 | 0/128
Serious Adverse Events (participants affected / at risk) | 0/128 | 0/128
Other Adverse Events (participants affected / at risk) | 0/128 | 0/128

LIMITATIONS AND CAVEATS:
Limitations of this trial include being conducted at a single site, being limited to those who are aged 17-25 years, and being limited to those who own smartphones or devices. Additional limitations include unpredictability of health coaches in terms of messaging patients on time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT04412954/Prot_SAP_000.pdf